CLINICAL TRIAL: NCT05216016
Title: Minnesota Retaining Employment and Talent After Injury/Illness Network Phase 2 RETAIN
Brief Title: Minnesota RETAIN Phase 2 (Sub-study)
Acronym: MN RETAIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Minnesota Department of Employment and Economic Development (Unknown); Minnesota Department of Labor and Industry (Unknown); Minnesota Department of Health (Other Government); Workforce Development, Inc. (Unknown); United States Department of Labor (Unknown); United States Social Security Administration (Unknown)
Responsible Party: Principal Investigator, Laura E. Breeher, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-006979; OD-36365-21-75-4-27 (Other Grant/Funding Number: Department of Labor and Social Security Administration)
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Injuries Related Work; Illness Related Work; Disability
Keywords: RETAIN; Minnesota RETAIN; MN RETAIN; Illness Recovery; Injury Recovery; Out of work help; Work placement assistance; Job help; Work Help; Help keeping my job; Stay at work; Return to work

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Individuals will receive a handout with additional job related services; e.g. Job Accommodation Network.
- Intervention Group (Experimental): Individuals will be assigned a dedicated Minnesota RETAIN Return-to-Work Case Manager. Intervention group participants will be referred for additional career and workforce development resources when needed.
  Interventions: Other: RETAIN Program
- Sub Study Group (Experimental): Individuals will be assigned a dedicated Minnesota RETAIN Return-to-Work Case Manager. Intervention group participants will be referred for additional career and workforce development resources when needed.
  Interventions: Other: RETAIN Program

INTERVENTIONS:
Other: RETAIN Program — Facilitates early intervention strategies to support workers in staying-at or returning-to-work (SAW/RTW) after injury or illness and preventing unnecessary disability. This is done by incorporating a Return-to-Work Case Manager as a member of the healthcare clinical team who acts as a liaison for the patient and assists in coordination of referrals between healthcare and Workforce Development services. Return-to-Work Case Managers will interact with treating providers of Minnesota RETAIN intervention group participants to ensure functionally based work restrictions are documented and shared with the patient's employer.
  Arms: Intervention Group; Sub Study Group

SUMMARY:
MN RETAIN Phase 2 Sub-study is a non-randomized trial to evaluate the impact of RETAIN program expansion and services on workforce retention and reduction of future workplace disability in the state of MN. The program is funded by US Department of Labor (US DOL) and sponsored jointly with the US Social Security Administration. There will be collaboration between partners to implement best practices in early intervention to support injured or ill employees in stay-at-work and return-to-work. MN RETAIN involves a partnership between Mayo Clinic and MN Department of Employment and Economic Development (DEED), MN Department of Labor and Industry (DLI), MN Department of Health (MDH), Workforce Development, Inc. (WDI), and the Governor's Workforce Development Board. MN DEED serves as the main recipient and administrator of the funding within the state with Mayo Clinic, DLI, and WDI, as subrecipients of the grant.

(Effective Date: 12/23/2021-05/16/2024) MN RETAIN Phase 2 : This study is a randomized control trial (RCT) to evaluate the impact of RETAIN program expansion and services on workforce retention and reduction of future workplace disability in the state of MN. The program is funded by US Department of Labor (US DOL) and sponsored jointly with the US Social Security Administration. There will be collaboration between partners to implement best practices in early intervention to support injured or ill employees in stay-at-work and return-to-work. MN RETAIN involves a partnership between Mayo Clinic and MN Department of Employment and Economic Development (DEED), MN Department of Labor and Industry (DLI), MN Department of Health (MDH), Workforce Development, Inc. (WDI), and the Governor's Workforce Development Board. MN DEED serves as the main recipient and administrator of the funding within the state with Mayo Clinic, DLI, and WDI, as subrecipients of the grant. During this Phase: additional collaborators: Mathematica Policy Research

ELIGIBILITY:
Inclusion Criteria

* > 18-years-old
* MN Resident
* Works in MN
* Employed at the time of enrollment
* Within 6 months of last day of work
* Meets one of the following:

  * Provider work restrictions of unable to work for at least 4 weeks
  * Per healthcare team anticipated to be unable to work for at least 4 weeks
  * Employer's inability to accommodate current work restrictions
* Meets one of the following:

  * Diagnosis of a work related or personal injury or illness that impacts employment
  * Invasive procedure (e.g., surgery) anticipated within the next 4-weeks that impacts employment
* Documentation of work restrictions (i.e., written note/form documentation in electronic medical record prior to enrollment)

Exclusion Criteria

* Legal representation/litigation at the time of enrollment related to a workers' compensation medical condition
* Does not have the capacity to give appropriate informed consent
* Employed by a RETAIN healthcare recipient or subrecipient with an existing return to work program for employees (i.e., Mayo Clinic employees)
* Workers' compensation recipients that have a qualified rehabilitation consultant (QRC) or a disability case manager (DCM)
* Pending application OR Receiving Social Security Disability Insurance (SSDI) or Supplemental Security Income (SSI)
* Self-Employed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5200 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Workers to maintain employment | 12 months
  Total number of workers employed at the time of program completion and who have maintained employment 12 months after enrollment.
Reduction on work disability at 1 years | 1 year
  Total number of enrollees that applied for SSDI or SSI during any of the 1 year after enrollment.
Reduction in long term work disability | 5 years
  Total number of enrollees that applied for SSDI or SSI during any of the 5 year after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Breeher, MD, MPH, Principal Investigator — Mayo Clinic; Clayton Cowl, MD,MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No